CLINICAL TRIAL: NCT02940067
Title: A Multimodal Approach to Improve Fitness and Surgical Outcomes for Patients Undergoing Pancreatic Resection
Brief Title: Enhancing Fitness Before Pancreatic Surgery
Acronym: MedEx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Surrey County Hospital NHS Foundation Trust (Other)
Collaborators: University of Surrey (Other)
Responsible Party: Principal Investigator, Jason George, Research Fellow, Royal Surrey County Hospital NHS Foundation Trust
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 197169
Record Dates: First submitted 2016-10-15; First posted 2016-10-20 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Pancreatic Cancer; Pancreatitis, Chronic
Keywords: prehabilitation; pancreatectomy; nutrition; exercise
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatitis, Chronic; Motor Activity | interventions — Preoperative Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MedEx (Experimental): This group will receive nutritional supplementation (based on components of the MEDiterranean diet) and supervised EXercise training for four weeks - hence the trial name, MedEx.
  Interventions: Other: MedEx
- Standard Care (No Intervention): This group will follow current standard preoperative care before scheduled pancreatic resection.

INTERVENTIONS:
Other: MedEx — A combination of dietary and exercise interventions over four weeks before scheduled pancreatic surgery
  Other Names: Prehabilitation
  Arms: MedEx

SUMMARY:
This is a pilot study to investigate the effect of prehabilitation on patients undergoing elective surgery for pancreatic disease.

DETAILED DESCRIPTION:
Pancreatic surgery is high risk. The injury associated with surgery causes a stress response, comprising a variety of hormonal and metabolic effects. Patients undergoing pancreatic surgery experience one of the largest stress responses. Prehabilitation is the process of enhancing an individual's fitness, thereby improving tolerance to an upcoming physiological stress such as surgery. Studies involving prehabilitation have been shown to improve recovery after surgery and reduce complication rates. There are currently no published reports of prehabilitation involving patients undergoing pancreatic surgery. This research study will explore the effect of prehabilitation in these patients.

Patients with pancreatic disease are some of the least fit surgical candidates due to the disease process. Exercise training can improve physical fitness before elective abdominal surgery and nutritional supplementation can also influence clinical course via different mechanisms. Patients with pancreatic disease are often malnourished for several reasons. We propose a multimodal approach to prehabilitation involving dietary and exercise interventions during a four-week period preceding elective surgery. Core data will be collected from cardiopulmonary exercise tests and blood tests (to assess insulin sensitivity), before and after prehabilitation. Secondary outcomes such as length of stay and complications will also be measured postoperatively.

ELIGIBILITY:
Inclusion Criteria:

Elective pancreatic resection

Exclusion Criteria:

Contraindication to cardiopulmonary exercise testing: unstable cardiac disease, lower limb dysfunction Emergency surgery Ischaemic ECG during cardiopulmonary exercise test Allergy to fish oil or olive oil

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2018-06-21 (Actual); Study Completion 2018-08-20 (Actual)

PRIMARY OUTCOMES:
Peak power - measured using cardiopulmonary exercise testing | Change in peak power between start and end of prehabilitation (4 weeks)
  cardiopulmonary fitness

SECONDARY OUTCOMES:
Insulin sensitivity - measured using the insulin clamp test | Change in insulin sensitivity between start and end of prehabilitation (4 weeks)
  insulin sensitivity
Length of stay | From date of operation until date of discharge
  Recovery
Complication rate | From date of operation until date of discharge
  Morbidity
Sleep | Change in sleep quality between start and end of prehabilitation (4 weeks)
  Sleep Quality
Fatigue | Change in fatigue levels between start and end of prehabilitation (4 weeks)
  Fatigue Levels
Well-being | Change in well-being scores between start and end of prehabilitation (4 weeks)
  Sense of Well-being

CONTACTS AND LOCATIONS:
Overall Officials: Tim Rockall, MD FRCS, Study Chair — MATTU, Royal Surrey County Hospital, Guildford, Surrey; Mike Scott, FRCA FFICM, Study Director — MATTU, Royal Surrey County Hospital, Guildford, Surrey; Jason George, MA MRCS, Principal Investigator — MATTU, Royal Surrey County Hospital, Guildford, Surrey; Martin Whyte, PhD FRCP, Study Director — University of Surrey, Guildford, Surrey; Joe Wainwright, BSc, Study Director — University of Surrey and Surrey Human Performance Institute
Locations (1):
- MATTU, Royal Surrey County Hospital, Guildford, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dunne DF, Jack S, Jones RP, Jones L, Lythgoe DT, Malik HZ, Poston GJ, Palmer DH, Fenwick SW. Randomized clinical trial of prehabilitation before planned liver resection. Br J Surg. 2016 Apr;103(5):504-12. doi: 10.1002/bjs.10096. Epub 2016 Feb 11. PMID 26864728
- [Background] Sato H, Carvalho G, Sato T, Lattermann R, Matsukawa T, Schricker T. The association of preoperative glycemic control, intraoperative insulin sensitivity, and outcomes after cardiac surgery. J Clin Endocrinol Metab. 2010 Sep;95(9):4338-44. doi: 10.1210/jc.2010-0135. Epub 2010 Jul 14. PMID 20631016
- [Background] Snowden CP, Prentis JM, Anderson HL, Roberts DR, Randles D, Renton M, Manas DM. Submaximal cardiopulmonary exercise testing predicts complications and hospital length of stay in patients undergoing major elective surgery. Ann Surg. 2010 Mar;251(3):535-41. doi: 10.1097/SLA.0b013e3181cf811d. PMID 20134313